CLINICAL TRIAL: NCT04434560
Title: A Phase II Trial of Surgery and Stereotactic Radiosurgery With Neoadjuvant Nivolumab and Ipilimumab in Patients With Surgically-resectable, Solid Tumor Brain Metastases
Brief Title: Neoadjuvant Immunotherapy in Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Sarah Sammons, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry); Duke University (Other)
Responsible Party: Sponsor-Investigator, Sarah Sammons, MD, Assistant Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103812; CA184-583 (Other: Bristol Myers Squibb)
Record Dates: First submitted 2020-06-12; First posted 2020-06-17 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Brain Metastases, Adult
Keywords: Pro00103812; Sammons; Non-small-cell lung carcinoma; Renal cell carcinoma; Urothelial carcinoma; Melanoma; Ovarian carcinoma; Triple negative breast cancer; Solid tumor; Brain metastases; Nivolumab; Ipilimumab; Opdivo; Yervoy
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Carcinoma, Transitional Cell; Melanoma; Ovarian Neoplasms; Triple Negative Breast Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (no neoadjuvant immunotherapy) (No Intervention): Patients will proceed to surgical resection with no nivolumab/ipilimumab given prior to surgery.
- Neoadjuvant Immunotherapy (Experimental): Patients will receive a single dose of neoadjuvant nivolumab and ipilimumab 7 days (± 3 days) prior to surgical resection.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab will be given at the FDA-approved dose of 3 mg/kg.
  Other Names: Opdivo
  Arms: Neoadjuvant Immunotherapy
Drug: Ipilimumab — Ipilimumab will be given at the FDA-approved dose of 1 mg/kg.
  Other Names: Yervoy
  Arms: Neoadjuvant Immunotherapy

SUMMARY:
The purpose of this phase 2 study is to assess the feasibility and efficacy of neoadjuvant immunotherapy in patients with previously untreated, surgically-resectable, solid tumor brain metastases. The primary objectives of this study are to 1) assess the feasibility of neoadjuvant ipilimumab and nivolumab treatment before surgery and stereotactic radiosurgery (SRS) in patients with solid tumor brain metastases as measured by the proportion of patients who have their surgery delayed or surgery never occurs, and 2) demonstrate that neoadjuvant immunotherapy will increase proliferation of circulating T-cells compared to baseline measurements. Exploratory objectives include describing patient progression free survival and overall survival, time to local and distant intracranial progression, and the rate of radiation necrosis. The rate of radionecrosis will also be explored, as immune expression profiles.

DETAILED DESCRIPTION:
Forty patients planned for standard of care resection of at least one solid tumor brain metastasis will be enrolled onto the study after providing informed consent. Primary tumor histology types are restricted to those known to extracranially respond to immunotherapy, and will include, but not be limited to, squamous non-small cell lung cancer (NSCLC), non-squamous NSCLC without known anaplastic lymphoma kinase (ALK), epidermal growth factor receptor (EGFR), and ROS mutation, renal cell carcinoma (RCC), melanoma, and triple negative breast cancer (TNBC) that is programmed death-ligand 1 positive (PD-L1 +). All participants will receive neoadjuvant immunotherapy and will receive a single infusion of nivolumab at a dose of 3 mg/kg and ipilimumab at a dose of 1 mg/kg 7 days (±3 days) prior to surgical resection of their metastases. Approximately three weeks after resection, patients in will then receive SRS per standard of care guidelines. Patients will be followed for 18 months after initiating study treatment. Up to 20 participants will be recruited and treated. Blood will be collected periodically during the study for correlative assessments.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must have at least 1 previously untreated, solid tumor brain metastases that are ≤4 cm in the largest direction. At least one of the metastases must be surgically resectable. All metastases must be planned for treatment with SRS. Primary tumor histology must be one of the following:

  1. Squamous NSCLC
  2. Non-squamous NSCLC without known ALK, EGFR, and ROS mutation
  3. RCC
  4. Urothelial carcinoma
  5. Ovarian carcinoma
  6. Melanoma
  7. Triple negative breast cancer that is PD-L1 positive
  8. Other solid tumor histologies may be eligible at the discretion of the PI if they are known to respond to immunotherapy containing regimens.
* 2. Patient must be asymptomatic or minimally symptomatic, requiring the equivalent of ≤ 4 mg dexamethasone daily for at least 7 days prior to enrollment
* 3. Patient or partner(s) meets one of the following criteria:

  1. Non-childbearing potential (i.e. not sexually active, physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile, or any male who has had a vasectomy). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Postmenopausal for purposes of this study is defined as 1 year without menses.; or
  2. Childbearing potential and agrees to use one of the following methods of birth control: approved hormonal contraceptives (e.g. birth control pills, patches, implants, or infusions), an intrauterine device, or a barrier method of contraception (e.g. a condom or diaphragm) used with spermicide.
* 4. Age ≥ 18 years of age at the time of entry into the study
* 5. Karnofsky Performance Score (KPS) ≥ 70
* 6. Prothrombin and Partial Thromboplastin Times ≤ 1.2 x normal prior to resection
* 7. Neutrophil count ≥ 1000 prior to resection
* 8. Hemoglobin ≥ 9 g/dl prior to resection
* 9. Platelet count ≥ 100,000/µl unsupported is necessary for eligibility on the study; however, because of risks of intracranial hemorrhage during resection, platelet count ≥ 125,000/µl is required for the patient to undergo resection, which can be attained with the help of platelet transfusion
* 10. Creatinine ≤ 1.5 x ULN (upper limit of normal) prior to resection
* 11. A signed informed consent form approved by the Institutional Review Board (IRB) will be required for patient enrollment into the study. Patients must be able to read and understand the informed consent document and must sign the informed consent indicating that they are aware of the investigational nature of this study
* 12. Ability to undergo MRI

Exclusion Criteria:

* 1. Females who are pregnant or breast-feeding
* 2. Patients with an impending, life-threatening cerebral herniation syndrome, based on the assessment of the study neurosurgeons or their designate
* 3. Patients with severe, active co-morbidity, defined as follow:

  1. Patients with an active infection requiring intravenous treatment or having an unexplained febrile illness (Tmax > 99.5°F/37.5°C)
  2. Patients with known immunosuppressive disease or known uncontrolled human immunodeficiency virus infection
  3. Patients with unstable or severe intercurrent medical conditions such as severe heart disease (New York Heart Association Class 3 or 4)
* 4. Patients who have not recovered from the toxic effects of prior chemo- and/or radiation therapy. Guidelines for this recovery period are dependent upon the specific therapeutic agent being used:
* 5. Patients must not have received immunotherapy within 3 months prior to enrollment
* 6. Patients with prior, unrelated malignancy requiring current active treatment in the last 3 years with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
* 7. Patients with a known history of hypersensitivity to nivolumab, or any components of nivolumab
* 8. Patients with a known history of hypersensitivity to ipilimumab, or any components of ipilimumab
* 9. Patients with active autoimmune disease requiring systemic immunomodulatory treatment within the past 3 months.
* 10. History and/or confirmed pneumonitis, or extensive bilateral lung disease on high resolution/spiral CT scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Sammons, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center — http://tischbraintumorcenter.duke.edu/
- See also: Duke Health — http://www.dukehealth.org/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In a Memo to File dated March 4, 2021, the removal of randomization in favor of a single-arm study in which all patients will receive neoadjuvant immunotherapy prior to their resection and SRS was proposed. One patient had already been randomized to receive standard of care surgery and SRS without neoadjuvant immunotherapy. This patient is not part of the analyses for the primary or secondary outcomes, as after the protocol amendment all patients were to receive neoadjuvant immunotherapy.
Period: Overall Study
Arm/Group | Standard of Care (no Neoadjuvant Immunotherapy) | Neoadjuvant Immunotherapy
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in the Neoadjuvant Immunotherapy group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (no Neoadjuvant Immunotherapy) | Neoadjuvant Immunotherapy | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Have Their Surgery Delayed by More Than 4 Days or Surgery Never Occurs as a Direct or Indirect Result of Ipilimumab and Nivolumab Treatment.
Time Frame: 10 days
Population: Outcome measure only applies to Neoadjuvant Immunotherapy; no participants were enrolled in the Neoadjuvant Immunotherapy group.
Arm/Group | Standard of Care (no Neoadjuvant Immunotherapy) | Neoadjuvant Immunotherapy
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Proliferation of Circulating T-cells as Measured by Mean Fold-change Between Baseline and Day 1 in Ki67 Levels.
Description: Ki-67 is a nuclear protein involved in cell proliferation regulation.
Time Frame: baseline to day 1
Population: as for outcome 1
Arm/Group | Standard of Care (no Neoadjuvant Immunotherapy) | Neoadjuvant Immunotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 10 days
Description: No participants were enrolled in the Neoadjuvant Immunotherapy group.
Arm/Group | Standard of Care (no Neoadjuvant Immunotherapy) | Neoadjuvant Immunotherapy
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (no Neoadjuvant Immunotherapy) (N=1) | Neoadjuvant Immunotherapy (N=0)
Pyramidal tract syndrome (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (no Neoadjuvant Immunotherapy) (N=1) | Neoadjuvant Immunotherapy (N=0)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Concentration impairment (Nervous system disorders) | 1 | 0
Dysphasia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Pyramidal tract syndrome (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT04434560/Prot_SAP_000.pdf